CLINICAL TRIAL: NCT04699357
Title: Shanghai Eye Disease Prevention and Treatment Center
Brief Title: The Effect and Safety of Different Doses of Atropine on Myopic Progression of Highly Myopic Children: Multi-centered Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SHDC12019111
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-01

CONDITIONS: High Myopia
MeSH Terms: interventions — Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): 0.01% atropine
  Interventions: Drug: Atropine
- Group 2 (Experimental): 0.04% atropine
  Interventions: Drug: Atropine
- Group 3 (Experimental): 0.1% atropine
  Interventions: Drug: Atropine

INTERVENTIONS:
Drug: Atropine — different concentrations (0.01%/0.04%/0.1%) of atropine were administered to high myopic children

SUMMARY:
Objective: to evaluate the efficacy of different concentrations of atropine eye drops in controlling the progression (diopter, axial length) of high myopia in young children, and to compare the compliance, adverse reaction and regression rate of different concentrations of atropine eye drops in myopia control.

Intervention: Group 1 (0.01% atropine group), Group 2 (0.04% atropine group), Group 3 (0.1% atropine group). During the 2-year intervention period after entering the group, each concentration of atropine eye drops were given every night at a fixed time before going to bed, one drop each time, implemented by parents (supervision), and the wechat small program was completed.

ELIGIBILITY:
Inclusion Criteria:

* The BCVA of distant vision is at least 0.5, near vision is at least 1.0, Titmus stereo vision is less than 80 seconds, far exotropia is less than 10 prism degrees, far esotropia is less than 6-8 prism degrees, and astigmatism is equal to or less than - 2.50 D;
* Myopia progressed more than 0.5D in the past year;
* Have normal thinking and language communication skills, and be able to actively cooperate with the treatment as required;
* Written informed consent of guardian and child.

Exclusion Criteria:

* Diseases of the study eye: keratitis, keratoconus, congenital cataract, glaucoma, fundus diseases; present situation with anterior segment or posterior segment inflammation, such as acute conjunctivitis, iridocyclitis;
* Systemic diseases affecting drug use: albinism, epilepsy, serious mental and neurological diseases, congenital heart disease, arrhythmia;
* Atropine allergy;
* Very low birth weight infants with birth weight less than 1500g;
* Receiving other treatment to control the development of myopia, including anticholinergic drugs such as atropine, or participated in other functional frame lens, multifocal soft lens in the past one year;
* Other situations that not suitable for participating in the trial as judged by the researcher

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 357 (Estimated)
Dates: Start 2021-07-04 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
changes of spherical equivalent | at least 3 years
  Spherical equivalent as measured by cycloplegia autorefraction
changes of axial length | at least 3 years
  AL was measured as the distance from the anterior corneal surface to the retinal pigment epithelium (RPE) using IOLMaster or Lenstar

CONTACTS AND LOCATIONS:
Overall Officials: Xun Xu, MD, Study Director — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (3):
- China (3):
  - Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai
  - Shanghai Ninth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided